CLINICAL TRIAL: NCT06229106
Title: Evaluation of the Symfony With Optiblue Intraocular Lens Compared to The Vivity IOL Under Mesopic Conditions
Brief Title: Symfony vs Vivity in Dim Light
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEP 23-001
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Symfony IOL (Active Comparator): The Symfony IOL is a lens designed to provide high quality vision up tp 26 inches reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
  Interventions: Device: Symfony IOL
- Vivity IOL (Active Comparator): The Vivity IOL is a lens that provides extended range of vision ranging from distance to near reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
  Interventions: Device: Vivity IOL

INTERVENTIONS:
Device: Symfony IOL — The Symfony IOL is a lens designed to provide high quality vision up tp 26 inches reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
  Arms: Symfony IOL
Device: Vivity IOL — The Vivity IOL is a lens that provides extended range of vision ranging from distance to near reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
  Arms: Vivity IOL

SUMMARY:
The purpose of this study is to evaluate the visual outcomes of the Symfony lens and the Vivity lens under mesopic lighting conditions in adult patients undergoing routine cataract surgery. Participants will be asked to read a visual acuity chart at different distances in dim light.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing bilateral lens extraction with implantation of an EDOF IOL with a target refraction of plano OU.
2. Gender: Males and Females.
3. Age: 50 years and older.
4. Willing and able to provide written informed consent for participation in the study
5. Willing and able to comply with scheduled visits and other study procedures.
6. Scheduled to undergo standard cataract surgery in both eyes, with 1 to 30 days between surgeries.
7. Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

1. Severe preoperative ocular pathology
2. Uncontrolled diabetes.
3. Use of any systemic or topical drug known to interfere with visual performance.
4. Contact lens use during the active treatment portion of the trial.
5. Any concurrent infectious/non-infectious conjunctivitis, keratitis, or uveitis.
6. Clinically significant corneal dystrophy.
7. Corneal irregularities potentially affecting visual acuity (i.e., keratoconus, corneal opacities.
8. History of chronic intraocular inflammation.
9. History of retinal detachment.
10. Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
11. Previous intraocular surgery.
12. Previous corneal refractive surgery (i.e., LASIK, PRK, RK).
13. Subject who declined any type of presbyopia correcting IOL due to concerns with visual disturbances (i.e., halos)
14. Previous keratoplasty
15. Severe dry eye
16. Pupil abnormalities
17. Subject who may reasonably be expected to require a secondary surgical intervention at any time during the study (other than YAG capsulotomy, i.e., LASIK)
18. Any clinically significant, serious, or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
19. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Sight, Sarasota, Florida
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Symfony Optiblue IOL: The Symfony IOL is a lens designed to provide high quality vision up tp 26 inches reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
  Symfony IOL: The Symfony IOL is a lens designed to provide high quality vision up tp 26 inches reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
- Clareon Vivity IOL: The Vivity IOL is a lens that provides extended range of vision ranging from distance to near reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
  Vivity IOL: The Vivity IOL is a lens that provides extended range of vision ranging from distance to near reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
Period: Overall Study
Arm/Group | Symfony Optiblue IOL | Clareon Vivity IOL
Started | 32 | 32
Completed | 31 | 31
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symfony Optiblue IOL | Clareon Vivity IOL | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.18 (7.02) | 70.16 (5.62) | 70.17 (6.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 17 | 17 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 30 | 30 | 60
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance Corrected Intermediate Visual Acuity at 66 cm Under Mesopic Conditions.
Description: logMAR visual acuity
Time Frame: 3 months after surgery
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Symfony Optiblue IOL: The Symfony IOL is a lens designed to provide high quality vision up to 26 inches reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
  Symfony IOL: The Symfony IOL is a lens designed to provide high quality vision up tp 26 inches reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
Arm/Group | Symfony Optiblue IOL | Clareon Vivity IOL
Number analyzed (Participants) | 31 | 31
logMAR | 0.27 (0.17) | 0.32 (0.11)

2. Secondary Outcome: Binocular Distance Corrected Intermediate Visual Acuity at 40 cm Under Mesopic Conditions.
Time Frame: 3 months after surgery
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Symfony Optiblue IOL: The Symfony IOL is a lens designed to provide high quality vision up to 26 inches reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
  Symfony IOL: The Symfony IOL is a lens designed to provide high quality vision up to 26 inches reducing the need for glasses after routine cataract surgery in patients with or without astigmatism.
Arm/Group | Symfony Optiblue IOL | Clareon Vivity IOL
Number analyzed (Participants) | 31 | 31
logMAR | 0.54 (0.15) | 0.52 (0.12)

3. Secondary Outcome: Binocular Low Contrast Distance Visual Acuity Under Mesopic Conditions
Description: Visual acuity measured at 4 m
Time Frame: 3 months after surgery
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Symfony Optiblue IOL | Clareon Vivity IOL
Number analyzed (Participants) | 31 | 31
logMAR | 0.44 (0.1) | 0.43 (0.1)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Symfony Optiblue IOL | Clareon Vivity IOL
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT06229106/Prot_SAP_000.pdf